CLINICAL TRIAL: NCT05407454
Title: Turkish Version of The Diabetes Quality of Life Brief Clinical Inventory Validity and Reliability
Status: Completed | Type: Observational
Sponsor: İlke KARA, PT (Other)
Collaborators: Bitlis Eren University (Other)
Responsible Party: Sponsor-Investigator, İlke KARA, PT, Co-Principal Investigator, Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Other Study IDs: BEU-21/11-1-E.1276
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes
Keywords: Diabetes; Quality of Life
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Patients with diabetes (all types)
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The original form of the Diabetes Quality of Life-Brief Clinical Inventory was first developed in 1999 to establish a valid and reliable form of diabetes-specific quality of life. Inventory items were developed to address the issues that have the greatest impact on assessing patient self-care behaviors and satisfaction with diabetes care. Items are ranked on a 5-point Likert scale and are in two general formats. One format includes satisfaction with treatment and quality of life and is scored from 1 (very satisfied) to 5 (not very satisfied). The second format includes the frequency of adverse effects of diabetes itself or diabetes treatment and offers response options from 1 (never) to 5 (always). Therefore, higher scores on the DQL-BCI items and subscales include negative values indicating problem frequency or dissatisfaction. In order to use the DQL scale more efficiently in clinics, Burroughs et al. organized the 15-item DQL-BCI in 2004.

SUMMARY:
This study aims to develop Turkish version of the Diabetes Quality of Life Brief Clinical Inventory (DQL-BCI) and to perform validity and reliability evaluations.

DETAILED DESCRIPTION:
The study will be carried out in two phases: DQL-BCI will be translated into Turkish and adapted to the cultural context, and the reliability and validity of the Turkish version of DQL-BCI will be investigated. The translation process will be performed in accordance with generally accepted international principles of translation and cultural adaptation of measurement tools. At least 150 subjects with type 2 diabetes will complete the Turkish version of DQL-BCI, the EQ-5D-3L questionnaire and the SF-12 quality of life questionnaire. The examination will provide information about the reliability and the construct validity of the studied tool.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-65 years old
* Diagnosed with diabetes for one year or more (Type 1 or Type 2)
* Literacy
* Being on at least one anti-diabetes medication

Exclusion Criteria:

* Not willing to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Aged between 18-65 years old with diabetes
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-08-07 (Actual)

PRIMARY OUTCOMES:
The Diabetes Quality of Life - Brief Clinical Inventory | 1 week
  The questionnaire consists of 15 questions, with no grouping into subscales or domains. Items are in two general formats. The first format is about the frequency of negative impacts of diabetes or odiabetes treatment and provides response options from "never" to "all the time". The second format is about the satisfaction with the treatment and QoL, and patients provide answers by selecting from "very satisfied" to "very dissatisfied". Answers to each question correspond to a score of 1-5, and 1 is the lowest score of a given parameter and 5 is the highest. The total score is the sum of scores of individual questions. The scoring ranges from 15 (the worst assessment of QoL) to 75 points (the best assessment of QoL).

CONTACTS AND LOCATIONS:
Locations (1):
- Bitlis Eren University, Bitlis, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No